CLINICAL TRIAL: NCT00810992
Title: Behavioral and Nutritional Therapy in Patients With Coronary Artery Disease According to Traditional Tibetan Medicine Protocol
Brief Title: Traditional Tibetan Medicine for Patients With Coronary Artery Disease
Acronym: TTM in CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Boris Bigalke, Prof. Dr., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 337/2008BO1 UKT
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease
Keywords: dietary, behavior; IDF criteria; coronary artery disease; Traditional Tibetan Medicine; coronary artery disease in patients, who have an increased cardiovascular risk profile according to the criteria by the International Diabetes Federation (IDF)
MeSH Terms: conditions — Coronary Artery Disease; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 Program A (Active Comparator): Recommendation for nutrition and behavior for patients with coronary artery disease according to the German Society of Nutritional Medicine and the International Task Force for the Prevention of Coronary Artery Disease
  Interventions: Behavioral: Nutritional and behavioral program A
- 2 Program B (Experimental): Recommendation for nutrition and behavior for patients with coronary artery disease according to the system of the Traditional Tibetan Medicine
  Interventions: Behavioral: Nutritional and behavioral program B

INTERVENTIONS:
Behavioral: Nutritional and behavioral program A — Recommendation for nutrition and behavior for patients with coronary artery disease according to the German Society of Nutritional Medicine and the International Task Force for the Prevention of Coronary Artery Disease
  Arms: 1 Program A
Behavioral: Nutritional and behavioral program B — Recommendation for nutrition and behavior for patients with coronary artery disease according to the system of the Traditional Tibetan Medicine
  Arms: 2 Program B

SUMMARY:
Coronary artery disease has a high death toll in the Western world. Changes in lifestyle, particularly in nutrition and physical activity may significantly reduce a severe coronary atherosclerosis within one year without the use of medication. Several dietary studies have shown that not only the progress of coronary artery disease can be slowed down, but it may also increase significantly the survival of these patients.

Up until now there is little known about therapeutic effects by complementary medicine. In particular, Traditional Tibetan medicine dietary programs have shown in few case reports that weight could be reduced in patients with obesity.

Therefore, the investigators developed a specific dietary program for patients with coronary artery disease, who have an increased cardiovascular risk profile according to the criteria by the International Diabetes Federation (IDF).

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* male and female
* coronary artery disease
* criteria of International Diabetes Federation (IDF)

Exclusion Criteria:

* <18 years old
* incapability for informed consent
* history of malignity, psychiatric disorder, tissue, thyroid gland and renal diseases, anorexia or bulimia
* administration of steroids or hormones
* pregnancy
* body mass index < 25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Body mass index | 6 months

SECONDARY OUTCOMES:
Intima media thickness HbA1C Lipid status Platelet activation markers as prognostic biomarkers | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

REFERENCES:
- [Background] Ornish D, Brown SE, Scherwitz LW, Billings JH, Armstrong WT, Ports TA, McLanahan SM, Kirkeeide RL, Brand RJ, Gould KL. Can lifestyle changes reverse coronary heart disease? The Lifestyle Heart Trial. Lancet. 1990 Jul 21;336(8708):129-33. doi: 10.1016/0140-6736(90)91656-u. PMID 1973470
- [Background] Singh RB, Dubnov G, Niaz MA, Ghosh S, Singh R, Rastogi SS, Manor O, Pella D, Berry EM. Effect of an Indo-Mediterranean diet on progression of coronary artery disease in high risk patients (Indo-Mediterranean Diet Heart Study): a randomised single-blind trial. Lancet. 2002 Nov 9;360(9344):1455-61. doi: 10.1016/S0140-6736(02)11472-3. PMID 12433513
- [Background] Michels KB, Wolk A. A prospective study of variety of healthy foods and mortality in women. Int J Epidemiol. 2002 Aug;31(4):847-54. doi: 10.1093/ije/31.4.847. PMID 12177033
- [Background] Trichopoulou A, Costacou T, Bamia C, Trichopoulos D. Adherence to a Mediterranean diet and survival in a Greek population. N Engl J Med. 2003 Jun 26;348(26):2599-608. doi: 10.1056/NEJMoa025039. PMID 12826634
- [Background] Bigalke B, Geisler T, Stellos K, Langer H, Daub K, Kremmer E, Seizer P, May AE, Lindemann S, Gawaz M. Platelet collagen receptor glycoprotein VI as a possible novel indicator for the acute coronary syndrome. Am Heart J. 2008 Jul;156(1):193-200. doi: 10.1016/j.ahj.2008.02.010. Epub 2008 Apr 23. PMID 18585516
- [Background] Bigalke B, Lindemann S, Ehlers R, Seizer P, Daub K, Langer H, Schonberger T, Kremmer E, Siegel-Axel D, May AE, Gawaz M. Expression of platelet collagen receptor glycoprotein VI is associated with acute coronary syndrome. Eur Heart J. 2006 Sep;27(18):2165-9. doi: 10.1093/eurheartj/ehl192. Epub 2006 Aug 21. PMID 16923742
- [Result] Liu L, Liu L, Ding Y, Huang Z, He B, Sun S, Zhao G, Zhang H, Miki T, Mizushima S, Ikeda K, Nara Y, Yamori Y. Ethnic and environmental differences in various markers of dietary intake and blood pressure among Chinese Han and three other minority peoples of China: results from the WHO Cardiovascular Diseases and Alimentary Comparison (CARDIAC) Study. Hypertens Res. 2001 May;24(3):315-22. doi: 10.1291/hypres.24.315. PMID 11409657
- [Derived] von Haehling S, Stellos K, Qusar N, Gawaz M, Bigalke B. Weight reduction in patients with coronary artery disease: comparison of Traditional Tibetan Medicine and Western diet. Int J Cardiol. 2013 Sep 30;168(2):1509-15. doi: 10.1016/j.ijcard.2013.07.034. Epub 2013 Jul 26. PMID 23890855
- See also: German Society of Nutritional Medicine — http://www.dgem.de
- See also: International Task Force for Prevention of Coronary Heart Disease — http://www.chd-taskforce.com/index_d.htm